CLINICAL TRIAL: NCT00822406
Title: Quantitative-Qualitative Clinical Trial to Evaluate the Effectiveness of Individualized Homeopathic Treatment in Perennial Allergic Rhinitis
Brief Title: Effectiveness of Individualized Homeopathic Treatment in Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Marcus Zulian Teixeira, Hospital das Clínicas da Universidade de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: marcus@homeozulian.med.br
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2009-01-27 (Estimated); Status verified 2009-01

CONDITIONS: Rhinitis
Keywords: allergy; rhinitis; homeopathy; double-blind
MeSH Terms: conditions — Rhinitis; Hypersensitivity | interventions — Homeopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): This arm received individualized homeopathic medicine during 6 months (initial phase), and completed three years (second phase)
  Interventions: Drug: homeopathic medicine
- 2 (Placebo Comparator): This arm received placebo during 6 months. After this period, all patients received individualized homeopathic medicine for three years.
  Interventions: Drug: homeopathic medicine; Drug: placebo

INTERVENTIONS:
Drug: homeopathic medicine — individualized homeopathic medicine
Drug: placebo — placebo - 6 months
  Arms: 2

SUMMARY:
A total of 41 adults with perennial allergic rhinitis were enrolled in a first double-blind placebo-controlled phase for six months, and treated on a weekly basis with sublingual doses of single individualized homeopathic medicines or placebo. After this closed initial phase, all patients were invited to participate in an long-term open-label controlled phase, in that they would receive homeopathic treatment for the maximum period of 36 months, and the results were compared with the improvement of initial phase. Signs and symptoms scores, rescue medication requirements and quality of life were assessed by questionnaires and personal clinical evaluation by a same independent researcher, before and after each phase. Primary and secondary clinical outcome were, respectively, specific and general allergic signs and symptoms scores. Total IgE titles were performed before and after each phase.

ELIGIBILITY:
Inclusion Criteria:

* moderate rhinitis
* to assign written informed consent

Exclusion Criteria:

* other chronic diseases
* corticosteroid use
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2002-07; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
specific allergic signs and symptoms score | 6 months

SECONDARY OUTCOMES:
general allergic symptoms score | 6 months

REFERENCES:
- [Derived] Teixeira MZ, Guedes CH, Barreto PV, Martins MA. The placebo effect and homeopathy. Homeopathy. 2010 Apr;99(2):119-29. doi: 10.1016/j.homp.2010.02.001. PMID 20471615